## **RESEARCH PROTOCOL (DAY 1)**



SK: researcher/PG 1
AAK: researcher/PG 2
EMA: researcher/PG 3



## **DAY 3**

SK to record clinical parameters & Check quality of temporary restorations

SK to examine and record clinical parameters

13) Apply Vaseline over GIC

14) Place patient under treatment pool

## **DAY 5,6 or 7**

EMA to give Questionnaire to parents/guardian AAK to check for quality of temporary restoration

1) Isolation with dental dam SK/PG 2) Disinfection with 30% Hydrogen Peroxide 3) Flush with 10% Iodine Tincture 4) Flush with 5% Thiosulphate 5) Remove Temporary GIC using Sterilized Round Bur **AAK** 6) Flush with sterilized saline 7) Paperpoint inserted into canal (2 paperpoints to be used each at 30s) 8) Canal preparation using sterilized K-File up to size 30 9) Flush with sterilized saline 10) Dry canals with Paperpoints 11) Placement of Vitapex using sterilized lentulospiral SK/EMA/AAK 12) Seal cavity with GIC restoration (Riva capsule)

## **Handling of sample**

